CLINICAL TRIAL: NCT02898311
Title: One-Tooth One-Time (1T1T) A Straightforward Approach to Replace Missing Teeth in the Posterior Region: a Case Series
Acronym: 1T1T
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Mainjot Amélie, Associate professor- Head of Clinic, University of Liege
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: TT001
Record Dates: First submitted 2016-08-27; First posted 2016-09-13 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Dental Implant Failed; Dental Prosthesis Failure
Keywords: CAD-CAM; composite dental resin; Immediate dental implant loading

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: immediate loading of posterior implants with chairside CAD-CAM composite crown

SUMMARY:
This study evaluates the success rate, as the biological and prosthesis complications, of posterior single-unit implants immediately loaded with a chair side Computer-Aided Design and Manufacturing (CAD-CAM) composite crown, after a follow-up period of 6 months,1,2,3,4 and 5 years.

Complementary ex vivo analyses will be performed to evaluate the wear of restorations. The time and cost benefit of the presented digital workflow, as patient centered outcomes will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

0 In good systemic health (ASA I/ II)

* Present with no contra indication against oral surgical interventions
* The tooth at the implant site(s) must have been extracted or lost at least 12 weeks before the date of implantation.
* At least 8 mm of bone in the vertical dimension
* At least 6 mm of bone in the bucco-lingual dimension.
* No need for bone augmentation procedure in any of the dimensions
* Full mouth plaque score (FMPI) lower or equal than 25%

Exclusion Criteria

* Autoimmune disease requiring medical treatment
* Medical conditions requiring prolonged use of steroids
* Use of Bisphosphonate intravenously or more then ˃ 3 years of oral use
* Infection (local or systemic) - patient with gingivitis or active local infection will undergo a medical treatment prior to his entrance to the study, each individual will be evaluated prior to study procedure for suitability, in case of systemic infection the evaluation will be based on medical anamneses, and if necessary will be referred to relevant medical tests.
* Current pregnancy or breastfeeding women
* Alcoholism or chronically drug abuse
* Immunocompromised patients
* Uncontrolled Diabetes
* Smokers
* Prisoners
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, or unreliability.

Local exclusion criteria:

* Sites treated with socket preservation techniques
* Untreated local inflammation
* Mucosal diseases or oral lesions
* History of local irradiation therapy in Head-Neck area
* Persistent intraoral infection (periodontitis, caries, …)
* Patients inadequate oral hygiene or unmotivated for normal home care.
* Removable prosthesis as an antagonist of the teeth to be replaced or absence of antagonistic teeth
* Severe bruxism or parafunctions

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2016-07; Primary Completion 2017-05 (Actual); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Implant complication rate | 6 months
Prosthesis complication rate | 6 months

SECONDARY OUTCOMES:
Evaluation of treatment duration, timing (in minutes) all the different steps of the surgical and prosthodontic procedure. | 1 day
Evaluation of patient satisfaction with VAS (visual analog scale) questionnaire | 1 day
Evaluation of patient satisfaction with VAS (visual analog scale) questionnaire | 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Liege University Hospital Center of Liege, Liège
  - University Hospital Center of Liège, Liège